CLINICAL TRIAL: NCT03782272
Title: Safety, Acceptability, and Feasibility of Enterade® in Children at Risk for Environmental Enteric Dysfunction in Kakamega County, Kenya
Brief Title: Safety, Acceptability, and Feasibility of Enterade®
Acronym: SAFE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study product bottles were found on site that did not meet product specifications. This prompted a 6-week safety review of participants (no study-related findings) and resulted in the study's termination.
Sponsor: PATH (Other)
Collaborators: Maseno University (Other); Kakamega County General Teaching & Referral Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1191395-1
Record Dates: First submitted 2018-05-16; First posted 2018-12-20 (Actual); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-07

CONDITIONS: Stunting; Environmental Enteric Dysfunction
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Intervention Model Description: This is a mixed-methods pilot study to assess the safety, acceptability, and feasible dosage of AA-ORS among children with mild to moderate stunting (LAZ between -1 and -3) who are at risk for EED and to assess the acceptability of this fluid supplementation for their caregivers. During the main study, up to 66 child participants will be randomized to receive 14 days of AA-ORS or placebo solution daily, dosing of up to 237 ml over a 3-hour period. Study staff and participants will be blinded to the study product allocation. Caregivers will store and return unused study product. Data collection methods to include direct observation of product consumption, structured surveys with caregivers, average daily volume consumed, and measurement of plasma/serum markers of metabolism, gut dysfunction, systemic inflammation, and micro-nutrient status pre- and post-administration of product.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AA-ORS (Experimental): Those receiving enterade oral re-hydration solution with amino acids
  Interventions: Dietary Supplement: Enterade
- Placebo (Placebo Comparator): Those receiving placebo solution without amino acids or rehydration salts
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Enterade — enterade® (an amino acid-based oral rehydration solution [AA-ORS]) is a medical food product that consists of oral rehydration salts, natural flavor, steviol (sweetener), purified water, and a blend of amino acids that drive the uptake of water and electrolytes.
  Arms: AA-ORS
Dietary Supplement: Placebo — a placebo solution containing natural flavor, steviol (sweetener), and purified water.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled pilot study to determine the safety, acceptability, and feasible pediatric dosage/tolerability of enterade® solution, an amino acid-based oral rehydration solution (AA-ORS), for potential use in the management of environmental enteric dysfunction (EED) among children aged 12-24 months in Kakamega County, Kenya.

Primary objectives:

1. To determine the safety of a 2-week course of AA-ORS among children with length-for-age Z-scores (LAZ) between -1 and -3.
2. To determine the feasibility and best tolerated dose of AA-ORS among children with LAZ between -3 and -1.

   Secondary objectives:
3. To determine the perceptions among caregivers on the acceptability of AA-ORS as a potential intervention for EED. (Qualitative)

   Exploratory objectives:
4. To determine the impact of AA-ORS on markers of metabolism, gut dysfunction, systemic inflammation, and micronutrient status among children with LAZ between -3 and - 1.

Qualitative results will not be reported on ClinicalTrials.gov.

DETAILED DESCRIPTION:
Environmental enteric dysfunction (EED) is an intestinal disorder common among people living in low-resource settings (LRS), which in children has been associated with increased risk of growth stunting, reduced cognitive development, and reduced oral vaccine responsiveness. An effective EED therapeutic would offer an opportunity to improve child growth and development in LRS. One promising intervention, enterade® (an amino acid-based oral rehydration solution [AA-ORS]), is a medical food product already sold in the United States. It consists of oral rehydration salts and a proprietary blend of amino acids designed to restore gut function, improve nutrient and electrolyte absorption, and improve barrier integrity. There is evidence that this AA-ORS reduces inflammation and promotes healing of damaged intestinal epithelium in murine models of intestinal damage (irradiated gut), and it may provide benefit to pediatric EED patients. Supplementation of amino acids may lessen or improve intestinal injury related to enteric illnesses commonly experienced in settings of poor hygiene and sanitation infrastructure. The results from this exploratory mixed-methods study could have broad implications for possible future studies among pediatric patients with intestinal injury resulting from EED and future product development and program strategies for EED interventions.

The study was terminated prematurely after study product was found on site that did not meet product specifications. Enrollment and all study product dosing was halted; previously enrolled participants were followed through planned study visits and assessments. An additional 6-week safety follow-up period was added to study procedures. No study-related adverse events were reported during per-protocol activities or from the additional 6-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

Pediatric and caregiver pairs (must meet inclusion criteria for both categories):

Child:

1. Is between 12 and 24 months of age.
2. LAZ between -3 and -1 standard deviations (SD).
3. At least one week post routine immunization, healthy child visit, or vitamin A supplementation visit at the study site.
4. Has a parent or legally acceptable representative willing and able to provide informed consent.
5. No plans for travel outside of the community for the duration of the study.

Caregiver of child:

1. Is a parent or legally accepted representative of a child eligible for this study.
2. Is 18 years of age or older.
3. Has a working mobile phone.
4. Is willing and able to provide informed consent.
5. If illiterate-there is at least one literate adult living in the child's household.

Exclusion Criteria:

Pediatric and caregiver pairs (must meet none of the exclusion criteria for either category):

Child:

1. Has any sign of acute illness, including but not limited to fever, cough, and diarrhea.
2. Is wasted (weight for length z-score < -2 or mid-upper arm circumference [MUAC] < 12.4 cm) or has pitting edema.
3. Is exclusively breastfed.
4. Is seeking medical attention at the health facility other than for routine, preventative care (e.g., immunization visit, vitamin supplementation).
5. Has suffered within the prior week from illnesses that might impact nutritional status (e.g., severe diarrhea or pneumonia; vomiting; persistent diarrhea; cleft lip or palate; blindness; tuberculosis; jaundice; renal or cardiac disease; cerebral palsy; known metabolic disorders; and chromosomal disorders, including trisomy 21).
6. Medical history of chronic health condition (i.e., HIV, hepatitis B or C, end stage renal disease, severe liver disease-absence of a diagnosis is sufficient).
7. Participating in any other clinical trials.
8. Recent (prior 2 weeks) use of antibiotics or any other medical treatments (including oral re-hydration solution), but not including vaccines or vitamin/mineral supplementation).
9. Cannot give the necessary biological (blood) sample.

Caregiver:

Reports diarrhea in the household in the prior 7 days.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kakamega County General Teaching and Referral Hospital, Kakamega, Kenya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AA-ORS | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AA-ORS | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Full Range); unit: months] | 18 [12 to 23] | 16 [13 to 21] | 18 [12 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kenya | 6 | 6 | 12
Length [Median (Full Range); unit: cm] | 78.95 [71.7 to 84.5] | 75.3 [71 to 79.3] | 78 [71.0 to 84.5]
Weight [Median (Full Range); unit: kg] | 10.55 [9.77 to 11.3] | 9.03 [8.5 to 10.5] | 10.0 [8.5 to 11.3]
Mid-upper arm circumference (MUAC) [Median (Full Range); unit: mm] | 150.5 [142 to 164] | 141 [138 to 150] | 145 [138 to 164]

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events or Serious Adverse Events
Description: Frequency of adverse events or serious adverse events in study product and placebo arms through 21 days of follow-up as assessed by physical/clinical examination.
Time Frame: 0-21 days
Population: This is the intention-to-treat population with all participants randomized and received at least one dose.
Measure: Count of Participants; unit: Participants
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 1 | 0

2. Primary Outcome: Volume of Daily Consumption of Study Product
Description: Total, average, and trends in daily study product volume consumed measured as milliliters per day through the 14 days of dosing.
Time Frame: 0-14 days
Population: Intention-to-treat
Measure: Median (Full Range); unit: ml
Groups:
- Pooled Arms: Due to study termination, insufficient data was collected for per-arm analysis. Only 2 participants completed the study per-protocol with a total of 12 having at least one dose of study product (target sample size was 66). Both AA-ORS and placebo arms data are pooled together.
Arm/Group | Pooled Arms
Number analyzed (Participants) | 12
ml | 212.5 [181 to 234]

3. Other Pre Specified Outcome: Exploratory - Metabolism: Plasma Concentration of Acylcarnitines
Description: Plasma concentration of acylcarnitines assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Exploratory - Gut Damage: Plasma Concentration of Intestinal Fatty Acid-binding Protein [I-FABP]
Description: Plasma concentration of intestinal fatty acid-binding protein [I-FABP] assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Exploratory - Microbial Translocation: Plasma Concentration of Soluble CD14 [sCD14]
Description: Plasma concentration of soluble CD14 [sCD14] assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Exploratory - Gut Repair: Plasma Concentration of Glucagon-like Peptide 2 [GLP-2]
Description: Plasma concentration of glucagon-like peptide 2 [GLP-2] assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Exploratory - Growth Hormone Axis: Plasma Concentration of Insulin-like Growth Factor 1 [IGF-1]
Description: Plasma concentration of insulin-like growth factor 1 [IGF-1] assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Exploratory - Growth Hormone Axis: Plasma Concentration of Fibroblast Growth Factor 21 [FGF21]
Description: Plasma concentration of fibroblast growth factor 21 [FGF21] assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Exploratory - Systemic Inflammation: Plasma Concentration of Alpha-1-acid Glycoprotein [AGP]
Description: Plasma concentration of alpha-1-acid glycoprotein [AGP] assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Exploratory - Systemic Inflammation:Plasma Concentration of C-reactive Protein [CRP]
Description: Plasma concentration of c-reactive protein [CRP] assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Exploratory - Micronutrient Status: Plasma Concentration of Ferritin
Description: Plasma concentration of ferritin assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Exploratory - Micronutrient Status: Plasma Concentration of Soluble Transferrin Receptor [sTfR]
Description: Plasma concentration of soluble transferrin receptor [sTfR] assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Exploratory - Micronutrient Status: Plasma Concentration of Retinol-binding Protein 4 [RBP4]
Description: Plasma concentration of retinol-binding protein 4 [RBP4] assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Exploratory - Micronutrient Status: Plasma Concentration of Thyroglobulin
Description: Plasma concentration of thyroglobulin assessed at baseline and day 15 of follow-up.
Time Frame: Day 0 and Day 15
Population: Due to study termination, exploratory analyses were not conducted on specimens collected.
Arm/Group | AA-ORS | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | AA-ORS | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA-ORS (N=6) | Placebo (N=6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT03782272/Prot_SAP_000.pdf